CLINICAL TRIAL: NCT02777346
Title: Evaluation of Emergency Suturing With Absorbable Versus Non-absorbable Suture Material in a Pediatric Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pediatric Clinical Research Platform (Other)
Responsible Party: Principal Investigator, Giorgio La Scala, PD, MD; Attending Surgeon, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: CER 09-057
Record Dates: First submitted 2016-05-17; First posted 2016-05-19 (Estimated); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Wounds and Injuries
Keywords: WOUNDS, PENETRATING; CHILD, PRESCHOOL; CHILD; INFANT; ADOLESCENT; SUTURES; POLYGLACTIN 910; POLYPROPYLENES
MeSH Terms: conditions — Wounds and Injuries; Wounds, Penetrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Absorbable (Experimental): Suture material: Polyglactin 910 thread (Vicryl Rapide®, Ethicon Inc).
  Interventions: Device: Absorbable
- Non Absorbable (Active Comparator): Suture material: Polypropylene thread (Prolene®, Ethicon Inc).
  Interventions: Device: Non absorbable

INTERVENTIONS:
Device: Absorbable — Wound suture by a resident physician. Two follow-up appointments (first at 4 to 21 days after the suture, according to the sutured site as defined by protocol, second at 6 months) Standardized photography of the wound before the suture and at the two subsequent follow-ups.
  Evaluation of the scar with a standardised form by a specialised nurse under medical supervision at the first follow-up and by a panel of investigators at 6 months using the pictures taken at the follow-up appointments.
  Arms: Absorbable
Device: Non absorbable — Wound suture by a resident physician. Two follow-up appointments (first at 4 to 21 days after the suture, according to the sutured site as defined by protocol, second at 6 months) Standardized photography of the wound before the suture and at the two subsequent follow-ups.
  Evaluation of the scar with a standardised form by a specialised nurse under medical supervision at the first follow-up and by a panel of investigators at 6 months using the pictures taken at the follow-up appointments.
  Arms: Non Absorbable

SUMMARY:
The investigators recruit patients admitted to the Pediatric Emergency Department of the Geneva's University Hospital with open wounds needing suture. The patients are treated with absorbable versus non-absorbable suture material according to randomization.

Outcomes are:

1. infection rate at the first follow-up (between 4 and 14 days, depending on the sutured site and defined by protocol)
2. scar appearance at a 6-months follow-up.

DETAILED DESCRIPTION:
The investigators recruit patients admitted to the Pediatric Emergency Department of the Geneva's University Hospital with open wounds needing suture. The patients are treated with absorbable versus non-absorbable suture material according to randomization.

After obtaining the patient's/parent's consent and randomization, the suture material will be provided.

Selection of the size of the thread and the date of the first follow-up are determined as follows:

* Face: Thread size 5-0 to 7-0, first follow-up 4-7 days
* Torso/back: Thread size 4-0 or 5-0, first follow-up 10-14 days
* Arms: Thread size 4-0 or 5-0, first follow-up 7- 10 days
* Hand: Thread size 5-0 or 6-0, first follow-up 7-10 days
* Legs: Thread size 4-0 or 5-0, first follow-up 7-14 days

The patients are examined by in the outpatient wound clinic by specialised nurses under medical supervision at the first follow-up, and at six months by one of the investigators.

Outcomes:

1. infection rate at the first follow-up (between 4 and 14 days, depending on the sutured site and defined by protocol)
2. scar appearance at a 6-months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient younger than 16 years of age with a wound requiring suture

Exclusion Criteria:

* Deep wounds with lesions of subcutaneous structures (tendons, nerves, etc.)
* Wounds with tissue loss
* Diabetic patients or patients treated with drugs potentially compromising cicatrization (e.g. steroids, immunosuppressors, etc.)
* Wounds caused by animal or human bites
* Sutures not performed in the emergency room
* Heavily soiled wounds

Ages: 1 Day to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 550 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Short-term infection risk | 4 to 21 days
  Scars classified as "no evidence of infection", "signs of inflammation" and "signs of active infection"

SECONDARY OUTCOMES:
Scar appearance | 6 months
  Scoring based on the Manchester scar scale

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio La Scala, MD PD, Study Director — University Hospital, Geneva
Locations (1):
- Geneva University Hospital, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No